CLINICAL TRIAL: NCT04724109
Title: Protocol for Study EQF01S: General Drug Use-Results Observational Study of Equfina® TABLETS 50 mg Observational Study on the Incidences of Adverse Drug Reactions in Patients With Parkinson's Disease (Including Patients With Hepatic Impairment)
Brief Title: A Study of Equfina® on the Incidences of Adverse Drug Reactions in Participants With Parkinson's Disease (Including Participants With Hepatic Impairment)
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: EQF01S
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Parkinsonian Disorders; Prospective; Non-interventional; Hepatic Impairment; Equfina
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Equfina: Participants with parkinson's disease will be administered Equfina 50 milligram (mg) tablets, orally, once daily in combination with levodopa-containing products. On the basis of symptoms, Equfina 100 mg tablet, orally, once daily may be selected for participants. All the participants will be observed for up to 24 weeks prospectively.
  Interventions: Drug: Equfina

INTERVENTIONS:
Drug: Equfina — Equfina oral tablets.

SUMMARY:
The purpose of the study is to investigate the incidences of psychiatric symptoms (example, hallucinations), somnolence and sudden onset of sleep, dyskinesia, and retinal degeneration-related events during treatment with Equfina in participants with parkinson's disease (including participants with hepatic impairment).

ELIGIBILITY:
Inclusion Criteria:

1. Participants with Parkinson's disease, who are naïve to Equfina

Exclusion Criteria:

1. Participants previously treated with Equfina
2. Participants who have contraindications on package insert of Equfina

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 1000 participants with parkinson's disease (including approximately 30 participants with hepatic impairment)
Sampling Method: Non-Probability Sample
Enrollment: 1088 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Adverse Drug Reactions (ADRs) | Up to 24 Weeks
  The numbers of participants based on the types of ADRs and AEs will be calculated. Number of participants with serious ADRs and serious AEs will be calculated. The numbers of participants based on the types of serious ADRs and serious AEs will be calculated.
Incidence Rate of ADRs Based on Baseline Characteristics of the Participants | Up to 24 Weeks
  Factors affecting safety will be investigated. Investigation for any association with various factors are to be performed employing appropriate analytical methods (example, logistic regression analysis). The factors include: gender, age, inpatient/outpatient status, duration of the disease, severity of Parkinson's disease (Hoehn and Yahr scale), presence/absence and details of psychiatric symptoms, severity of hepatic impairment, comorbidities, presence/absence of surgical treatment for Parkinson's disease, presence/absence of comorbid retinal pathology, history of drug allergy, presence/absence of pregnancy/breast-feeding (for females only), and history of smoking.
Change From Baseline in Symptoms of Parkinson's Disease After the Start of Treatment with Equfina | Baseline, up to Week 24
  Parkinson's disease motor examination will be performed using Unified Parkinson's Disease Rating Scale (UPDRS) part III, motor signs of parkinson's disease during "ON" time will be evaluated. It contains following items: (1) speech, (2) facial expression, (3) tremor at rest, (4) action or postural tremor of hands, (5) rigidity, (6) finger taps, (7) hand movements, (8) pronation-supinational movements of hands, (9) leg agility, (9) arising from chair, (10) posture, (11) gait, (12) postural stability, (13) body bradykinesia and hypokinesia. Each item is rated on a 5-point likert scale of 0 to 4: 0=normal, 1=slight, 2=mild, 3=moderate, and 4=severe. Higher the score the greater will be the severity.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Eisai Trial Site 2, Osaka
  - Eisai Trial Site 1, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.